CLINICAL TRIAL: NCT04297592
Title: Antibiotic Prophylaxis in High-Risk Arthroplasty Patients
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nicholas A. Bedard, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-001273
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Infections Joint Prosthetic; Overweight or Obesity; MSSA Colonization; MRSA; Chronic Kidney Diseases; Diabetes; Autoimmune Diseases; Inflammatory Disease; Tobacco Use
Keywords: total hip arthroplasty; total knee arthroplasty; hip replacement; knee replacement; periprosthetic joint infection; prophylaxis; antibiotics
MeSH Terms: conditions — Overweight; Obesity; Renal Insufficiency, Chronic; Diabetes Mellitus; Autoimmune Diseases; Tobacco Use | interventions — Cephalexin; Doxycycline; Cefadroxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Additional Antibiotic Group (Active Comparator): Patients will receive an oral antibiotic to be started after completion of standard perioperative antibiotics following primary hip or knee arthroplasty. Oral antibiotic will either be a first-generation cephalosporin (Cefadroxil or Cephalexin) or Doxycycline based upon patient allergies, kidney function and result of nasal colonization testing for MRSA.
  Interventions: Drug: Cephalexin; Drug: Doxycycline; Drug: Cefadroxil
- Control Group - No Additional Antibiotic (No Intervention): Patients will receive standard perioperative antibiotics following primary hip or knee arthroplasty and no additional antibiotics.

INTERVENTIONS:
Drug: Cephalexin — 500 mg oral tablet, 4 times daily for 7 days
  Other Names: Keflex
  Arms: Additional Antibiotic Group
Drug: Doxycycline — 100 mg oral tablet, 2 times daily for 7 days
  Arms: Additional Antibiotic Group
Drug: Cefadroxil — 500 mg oral tablet, 2 times daily for 7 days
  Other Names: Duricef
  Arms: Additional Antibiotic Group

SUMMARY:
To determine the effectiveness of a 7-day course of an oral, prophylactic antibiotic on the incidence of periprosthetic joint infection and wound complications following primary total hip and knee arthroplasty in a high-risk patient population.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate whether a 7-day course of an oral, prophylactic antibiotic following elective, primary total hip and knee arthroplasty effectively decreases the risk of periprosthetic joint infection or wound complications following surgery in a patient population that is high-risk for these complications. Patient with one or more of the following risk factors are considered high-risk for periprosthetic joint infection and/or wound complications: body mass index over 35kg/m^2, diagnosis of diabetes, chronic kidney disease, active tobacco user, nasal colonization of methicillin-resistant Staphylococcus aureus and/or methicillin-sensitive Staphylococcus aureus, or autoimmune/inflammatory disease.

Study participants will be randomized to either a 7-day course of an oral, prophylactic antibiotic following surgery or no additional antibiotic. All other standard perioperative total joint arthroplasty care will remain the same for both groups, including 24-hours of perioperative antibiotics. Outcomes assessed will include surgical wound complications occurring within 90-day of surgery and periprosthetic joint infection occurring within 90-day and 1-year of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for elective, primary total hip arthroplasties (THA) or total knee arthroplasties (TKA).
* Patient is considered high-risk for developing Periprosthetic joint infections (PJI) based on having at least one of the following criteria:
* Body mass index (BMI) > 35 kg/m^2;
* Diagnosis of diabetes mellitus;
* Active tobacco smoker;
* Chronic kidney disease;
* Autoimmune disease;
* Nasal colonization with methicillin-resistant Staphylococcus aureus (MRSA) or methicillin-sensitive Staphylococcus aureus (MSSA).

Exclusion Criteria:

* Inability to consume oral antibiotics.
* Allergy to antibiotic alternatives in the protocol.
* History of clostridium difficile colitis.
* Revision hip or knee arthroplasty procedure.
* Non-elective surgery.
* Hemiarthroplasty.
* Unicompartmental knee arthroplasty.
* Simultaneous bilateral THA or TKA.
* Will have subsequent THA or TKA within 12 weeks of the index study procedure.
* Pregnant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4618 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Periprosthetic joint infections | Within 90-days primary hip or knee arthroplasty
  Defined by Musculoskeletal Infection Society (MSIS) criteria
Periprosthetic joint infections | Within 1-year of primary hip or knee arthroplasty
  Defined by Musculoskeletal Infection Society (MSIS) criteria

SECONDARY OUTCOMES:
Wound complication | Within 90 days of primary hip or knee arthroplasty
  Defined by at least one of the following: surgical wound dehiscence, skin necrosis at the surgical site, persistent surgical wound drainage (fluid extrusion from the operative site occurring beyond 72 hours from index surgery), superficial surgical site infection treated with new prescription of antibiotics or a change in study antibiotics but not meeting criteria for periprosthetic joint infection.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Bedard, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inabathula A, Dilley JE, Ziemba-Davis M, Warth LC, Azzam KA, Ireland PH, Meneghini RM. Extended Oral Antibiotic Prophylaxis in High-Risk Patients Substantially Reduces Primary Total Hip and Knee Arthroplasty 90-Day Infection Rate. J Bone Joint Surg Am. 2018 Dec 19;100(24):2103-2109. doi: 10.2106/JBJS.17.01485. PMID 30562290
- [Background] Li B, Webster TJ. Bacteria antibiotic resistance: New challenges and opportunities for implant-associated orthopedic infections. J Orthop Res. 2018 Jan;36(1):22-32. doi: 10.1002/jor.23656. Epub 2017 Aug 11. PMID 28722231
- [Background] Kurtz SM, Lau E, Watson H, Schmier JK, Parvizi J. Economic burden of periprosthetic joint infection in the United States. J Arthroplasty. 2012 Sep;27(8 Suppl):61-5.e1. doi: 10.1016/j.arth.2012.02.022. Epub 2012 May 2. PMID 22554729